CLINICAL TRIAL: NCT02493621
Title: Compare Effectiveness of Epidural vs. Lumbar Plexus Blocks in Total Hip Arthroplasty (THA) Patients Using Multimodal Pain Control
Brief Title: Compare Epidural vs. Lumbar Plexus Analgesia After Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sylvia Wilson, Associate Professor, Medical University of South Carolina
Other Study IDs: Pro00040998
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-06

CONDITIONS: Arthropathy of Hip
Keywords: Pain, Postoperative; Nerve Block; Anesthesia, Epidural
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lumbar plexus: Patients received a preoperative lumbar plexus nerve block (20 ml, ropivacaine 0.5%) for postoperative pain management.
- Lumbar Epidural: Patients received a lumbar epidural preoperatively for postoperative pain management. Epidural infusions of ropivacaine 0.2% were initiated intraoperatively, administered until the morning of postoperative day 1, and titrated to patient comfort.

SUMMARY:
The goal of this retrospective chart review is to evaluate if the implementation of lumbar plexus block placement for postoperative pain have improved conditions in the postoperative period for patients undergoing total hip arthroplasty when compared to the placement of epidurals for postoperative pain management.

DETAILED DESCRIPTION:
Primary outcome: 48 hour opiate consumption in patients following THA. ' Secondary outcome: Time to first ambulation, assistance needed with ambulation, opiate and regional related side effects, time to discharge orders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosis of:

  1. Primary THA, (identified by CPT code 27130)
  2. Either a) Epidural (CPT code 62319) or b) Lumbar plexus peripheral nerve block (CPT 62311 or 64449)
* Perioperative multimodal medication
* Hospitalized from July 1, 2012 to December 17, 2014.

Exclusion Criteria:

* THA Revision
* ICU admission postoperatively
* History of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study team will identify subject by the Primary Diagnosis of THA, (identified by CPT code 27130) and 2) either a) Epidural (CPT code 62319) or b) Lumbar plexus peripheral nerve block (CPT 62311 or 64449) with the administration of multimodal medication.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria included primary, elective THA with either lumbar epidural (n=547) or lumbar plexus peripheral nerve block (n=219) for postoperative analgesia. Exclusion criteria included THA revision, traumatic fractures, non-elective surgeries, and postoperative ICU admission. 342 epidural &107 lumbar plexus patients met inclusion criteria.
Pre-assignment Details: Subjects meeting inclusion criteria were assigned a chronological number based on the date of their operation (Epidural 1-342; Lumbar plexus 1-107) and then randomized using Microsoft Excel. Data were collected on the first 58 randomized subjects in each group; 58 epidural patients and 58 lumbar plexus patients.
Period: Overall Study
Arm/Group | Lumbar Plexus | Lumbar Epidural
Started | 58 | 58
Completed | 58 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumbar Plexus | Lumbar Epidural | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (4.50) | 61.3 (1.99) | 60.8 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 64
  Male | 23 | 29 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 47 | 45 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Opiate Consumption
Description: Cumulative opiate consumption in intravenous (IV) morphine mg equivalents (MME)
Time Frame: 48 hours postoperative
Measure: Mean (Standard Error); unit: Opiate Consumption (IV MME)
Arm/Group | Lumbar Plexus | Lumbar Epidural
Number analyzed (Participants) | 58 | 58
Opiate Consumption (IV MME) | 64.8 (3.32) | 81.3 (4.13)

2. Secondary Outcome: Time of First Ambulation
Description: Time of first ambulation relative to anesthesia end time (hours)
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Lumbar Plexus | Lumbar Epidural
Number analyzed (Participants) | 58 | 58
Hours | 24.6 (2.01) | 31.7 (1.54)

ADVERSE EVENTS:
Arm/Group | Lumbar Plexus | Lumbar Epidural
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No